CLINICAL TRIAL: NCT05180422
Title: A Phase I/II Study of AMG 510 in Combination With MVASI in Patients With Advanced, Unresectable or Metastatic KRAS G12C Mutant NSCLC With Asymptomatic Brain Metastasis.
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: Criterium, Inc. (Industry)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 02AT21-KRAS
Record Dates: First submitted 2021-12-06; First posted 2022-01-06 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — sotorasib; Bevacizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dose Expansion (Experimental): AMG 510/MVASI
  Interventions: Drug: AMG 510; Drug: MVASI

INTERVENTIONS:
Drug: AMG 510 — Continuous once daily (QD) oral dosing (Days 1-21 each cycle) with or without food.
Drug: MVASI — Intravenous (i.v.) infusion every 21 days (i.e. Day 1 of each 21-day cycle).

SUMMARY:
This is a multicenter, non-randomized, open-label, phase I/II study to evaluate the safety and tolerability of AMG 510 plus MVASI in subjects with advanced KRAS p.G12C mutant non-small cell lung cancer (NSCLC) with small, untreated brain metastases.

DETAILED DESCRIPTION:
Each patient is scheduled to receive AMG 510 (KRASG12C inhibitor) in combination with MVASI (vascular endothelial growth factor [VEGF] inhibitor; bevacizumab biosimilar); both drugs will be provided by the study:

AMG 510:

Continuous once daily (QD) oral dosing (Days 1-21 each cycle) with or without food.

MVASI:

Intravenous (i.v.) infusion every 21 days (i.e. Day 1 of each 21-day cycle).

The study will be conducted in 2 parts. The dose expansion part of the study (Part 2) can open once the maximum tolerated dose (MTD) and/or a biologically active dose (e.g. recommended phase 2 dose [RP2D]) using a 3+3 study design has been determined in Part 1.

CNS response will be assessed using RANO-BM criteria, and non-CNS objective response will be based on Solid Tumor Response Criteria [RECIST v1.1] assessment of overall tumor burden at baseline versus that detected on subsequent CT/MRI re-scans. This includes a brain MRI on C2D1 (21 days) and a CT chest/abdomen/pelvis (C/A/P) at 6 weeks, then brain MRI at 15 weeks and CT C/A/P imaging at 12-16 weeks, and then every 4 cycles (every 12 weeks) while on study. It is intended that patients will be treated until disease progression or intolerable toxicity. Patients will be followed for survival for up to 18 months after ending study treatment.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all of the following inclusion criteria to be eligible for enrollment into the study:

1. Signed and dated written informed consent.
2. Male or female ≥ 18 years of age at the time of informed consent.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2.
4. As estimated by study physician, life expectancy ≥ 12 weeks.
5. Histologically proven, locally advanced, recurrent or metastatic KRAS G12C mutant non-small cell lung cancer (NSCLC), with pathological documentation of KRAS p.G12C mutation identified through DNA sequencing either in tumor tissue or blood circulating tumor DNA.
6. At least one untreated brain metastasis ≥ 5mm in diameter in any line of treatment:

   * Subjects with largest measurable intracranial lesion ≥5 mm but <10 mm may be allowed to enroll upon agreement with investigator (for patients with target lesions of ≥ 5mm but <10 mm, 1.5 mm slice thickness brain MRI is required).
   * "Untreated" refers to the lesion not being previously treated with stereotactic radiosurgery (SRS).
   * Prior treatment with whole brain radiation therapy or local surgery is permissible provided unequivocal progression in the lesion has since occurred and completion 14 days prior to study enrollment.
7. For at least 7 days prior to first dose of AMG 510 and MVASI in this study: Patient must be asymptomatic from CNS metastases and on a stable dose of corticosteroids.
8. Able to take oral medications and willing to record daily adherence to investigational product.
9. As assessed by electrocardiogram (ECG) completed ≤ 14 days before initiation of protocol treatment, the corrected QT interval (QTc) will be calculated by Fridericia's method (QTcF) - see Section 7.12. Eligible candidates (male or female) must have the following QTcF value on baseline ECG:

   • QTcF ≤ 470 ms.

   The average QTcF value from three (3) separate ECG tracings, each performed on the same day (ideally at least 5 minutes apart), will serve as the baseline QTcF value used to meet eligibility.
10. Adequate organ and bone marrow function resulted ≤ 14 days prior to first dose of protocol-indicated treatment:

    1. Prothrombin time (PT) and partial thromboplastin time (PTT) < 1.5x institutional upper limit of normal (ULN).
    2. Absolute neutrophil count (ANC) > 1500/µL.
    3. Hemoglobin ≥ 9 g/dL.
    4. Platelets ≥ 75,000/µL.
    5. Total bilirubin ≤ 1.5x ULN; or

       * < 2x ULN in subjects with documented Gilbert's syndrome; or
       * < 3x ULN in subjects for whom the indirect bilirubin level suggests an extrahepatic source of total bilirubin elevation).
    6. AST (SGOT) and ALT (SGPT) ≤ 2.5x ULN; or

       • ≤ 5x ULN if liver metastases are present.
    7. Serum creatinine ≤ 1.5mg/dL.
11. Women must not be breastfeeding and further agree to not breastfeed during study treatment; and for at least 1 week (7 days) after patient's final dose of AMG 510, and for at least 6 months (183 days) after patient's final dose of MVASI.
12. A woman of childbearing potential (WOCBP) - see Appendix 3 for definition of WOCBP - must have a negative serum or urine β-hCG pregnancy test (or in cases of β-hCG tumor production, may be confirmed not pregnant by uterine ultrasound during screening) within 14 days prior to receiving first dose of protocol-indicated treatment to be eligible, and must agree to follow instructions for using acceptable contraception (Appendix 3) from the time of signing consent, and until at least 6 months (183 days) after her final dose of AMG 510 and MVASI.
13. A man able to father children (see Appendix 3 for definition) who is sexually active with a WOCBP must agree to follow instructions for using acceptable contraception (Appendix 3), from the time of signing consent, and until at least 6 months (183 days) after his final dose of AMG 510 and MVASI.

Exclusion Criteria:

Patients meeting any of the following criteria will not be permitted to enter the trial:

1. Other coexisting malignancies or malignancies diagnosed within the previous 2 years are not eligible.

   * Exceptions to this include non-melanoma skin cancer, cervical cancer in-situ, well-differentiated thyroid cancer or prostate cancer.
   * Other cancers that per assessment of the principal investigator are not prognosis-limiting can be allowed after review by the principal investigator. If there is no evidence of disease for at least 3 years prior to initiating treatment in this study, patients may be eligible.
2. Prior receipt of AMG-510, other KRAS G12C inhibitors, or VEGF inhibitors for the treatment of non-small cell lung cancer.
3. Myocardial infarction within 6 months of study Day 1, symptomatic congestive heart failure equivalent to New York Heart Association > Class II (see Appendix 2) or unstable (requiring hospitalization or heart catheterization) angina currently.
4. Patient on full dose, therapeutic anticoagulation for thromboembolic event, arrhythmia, or prothesis with coumadin.
5. Evidence of clinically significant hemorrhage (per study physician) in untreated CNS lesion(s) on screening MRI.
6. Major surgery within 28 days of enrollment or presence of a non-healing wound.
7. Proteinuria of greater than 1 gram per 24 hours.
8. Recent history of moderate or severe hemoptysis within 7 days (greater than 20mL of pure blood within 24 hours).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-06-15 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Dose Exploration | 21 days
  To determine the feasibility and safety of AMG 510 in combination with MVASI for the treatment of patients with KRAS G12C mutant NSCLC with asymptomatic, untreated brain metastases.
  For patients enrolled in the dose exploration part of the study (anticipated to be the initial 9-18 patients participating in the study), whose participation will establish the recommended phase 2 dose (RP2D), dedicated surveillance and expedited reporting of Dose Limiting Toxicity (DLT) required for 21 days after initiating protocol-indicated treatment. Satisfactory completion of the physical exam and safety labs is required to help detect evidence of past or present DLT as having occurred during the first 21 days of protocol-indicated treatment.
Dose Expansion | 18 weeks
  To determine the CNS objective response and rate of salvage radiation to the CNS 18 weeks after therapy initiation.
  The CNS objective response rate using Rando-BM will be evaluated at 18 weeks. Whether or not the patient requires salvage radiation therapy will be evaluated at 18 weeks
Dose Exploration | 21 days
  Safety and tolerability (phase I component).
  Dedicated surveillance and expedited reporting of Dose Limiting Toxicity (DLT) is required for 21 days after initiating protocol-indicated treatment A minimum of 6 patients will be treated at the Maximum tolerated dose on the phase I portion of the study in order to obtain sufficient toxicity data prior to proceeding to the phase II evaluation of this regimen
Dose Expansion | 18 weeks
  CNS objective response, assessed using RANO-BM.
Dose Expansion | 18 weeks
  Initiation of salvage radiation therapy to the CNS at 18 weeks (phase II component).

SECONDARY OUTCOMES:
Dose Expansion | 18.5 months
  To evaluate systemic disease control by progression free survival and overall survival.
Dose Expansion | 18 weeks
  Non-CNS overall response (ORR), assessed using RECIST v1.1.
Dose Expansion | 18.5 months
  Non-CNS progression-free survival (PFS).
Dose Expansion | 18.5 months
  Overall Survival (OS).

CONTACTS AND LOCATIONS:
Overall Officials: Wade Iams, MD, MSCI, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt Ingram Cancer Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No